CLINICAL TRIAL: NCT00825474
Title: A Prospective Randomized Trial Comparing Partial Hepatectomy and TACE Plus PEI for Small Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospotal, Eastern Hepatobiliary Surgery Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EHBH-RCT-2008-003
Record Dates: First submitted 2009-01-15; First posted 2009-01-21 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: small hepatocellular carcinoma; partial hepatectomy; TACE plus PEI
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- survival rate (Experimental): therapeutic effect of partial hepatectomy or TACE plus PEI for small hepatocellular carcinoma
  Interventions: Other: operation;TACE plus PEI

INTERVENTIONS:
Other: operation;TACE plus PEI — Under normal rules, the operation group open abdomen to perform operation through subtotal incision while the patient has been general anesthesia with trachea cannula. The operation range on hepatic tissue of un-tumor tissue around tumor should maintain at least 1cm. As for the micro-create treatment combination group, taking TACE all through arteria cruralies super-elect arteria hepatica and injecting MITO、FUDR、iodipin. By B transonogram guiding to nyxis liver biopsy,and perform per cutem absolute alcohol injection treatment.
  Other Names: surgical resection

SUMMARY:
Presently,the diagnostic method of small hepatocellular carcinoma has been greatly elevated in China.The treatment is being from simplification to diversification,from entirety to individualization.Confronting small hepatocellular carcinoma,we not select simple operation treatment but select a treatment that have more predominance and more fitting with patients in various kinds of treatment methods;including operation ,TACE,PEI,et al.which is better ? There are many arguments.

DETAILED DESCRIPTION:
randomly put in group standard:

1. via clinical diagnosis and confirm it is primary liver cancer, and not accept any anticancer treatment.
2. age: 18-70 years.
3. early hepatocyte cancer，which is single focus of infection diameter ≤ 3 cm.
4. estimate tumor can gain treatment of curing operation or TACE plus PEI.
5. better liver function (Child-Pugh，class A or B).

Case loads: 160 residents with small hepatocellular carcinoma in China

Therapeutic regimen: under normal rules, the operation group open abdomen to perform operation through subtotal incision while the patient has been general anesthesia with trachea cannula. The operation range on hepatic tissue of un-tumor tissue around tumor should maintain at least 1cm. As for the micro-create treatment combination group, taking TACE all through arteria cruralies super-elect arteria hepatica and injecting MITO、FUDR、iodipin. By B transonogram guiding to nyxis liver biopsy,and perform per cutem absolute alcohol injection treatment.

Research end-point:

1. ensemble life span.To compare 1、2 and 3 year overall survival rate in hepatectomy and TACE plus PEI for small hepatocellular carcinoma
2. intraliver recurrence rate; distant metastasis rate; non-tumor life span; band tumor life span

Telephone call at any time

ELIGIBILITY:
Inclusion Criteria:

1. via clinical diagnosis and confirm it is primary liver cancer, and not accept any anticancer treatment.
2. age:18-70years
3. early hepatocyte cancer，which is single focus of infection diameter ≤3cm.
4. estimate tumor can gain treatment of curing operation or micro-create treatment combineation
5. better liver function (Child-Pugh，class A or B)

Exclusion Criteria:

1. reject to attend；
2. impossible to come to our hospital for physical examination regularly.
3. cancer epitome、seed focus、lymph node or distant metastasis
4. Blood clotting function hindrance;
5. serious heart、lung、kidney disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2008-08; Primary Completion 2009-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
overall survival | 2010

CONTACTS AND LOCATIONS:
Overall Officials: shen feng, MD, Study Chair — Eastern Hepatobiliary Surgery Hospital
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality, China